CLINICAL TRIAL: NCT00698230
Title: Randomized Study to Evaluate the Safety and Efficacy of INCB013739 Plus Metformin Compared to Metformin Alone on Glycemic Control in Type 2 Diabetic Subjects
Brief Title: Safety and Efficacy of INCB013739 Plus Metformin Compared to Metformin Alone on Glycemic Control in Type 2 Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 13739-202
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A - INCB013739 & Metformin (Experimental): INCB013739 5 mg QD and Metformin
  Interventions: Drug: INCB013739; Drug: Metformin
- Treatment B - INCB013739 & Metformin (Experimental): INCB013739 15 mg QD and Metformin
  Interventions: Drug: INCB013739; Drug: Metformin
- Treatment C - INCB013739 & Metformin (Experimental): INCB013739 50 mg QD and Metformin
  Interventions: Drug: INCB013739; Drug: Metformin
- Treatment D - INCB013739 & Metformin (Experimental): INCB013739 100 mg QD and Metformin
  Interventions: Drug: INCB013739; Drug: Metformin
- Treatment E - INCB013739 & Metformin (Experimental): INCB013739 200 mg QD and Metformin
  Interventions: Drug: INCB013739; Drug: Metformin
- Treatment F - Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo comparator matching INCB013739

INTERVENTIONS:
Drug: INCB013739 — INCB013739 5 mg QD tablet
  Arms: Treatment A - INCB013739 & Metformin
Drug: INCB013739 — INCB013739 15 mg QD tablet
  Arms: Treatment B - INCB013739 & Metformin
Drug: INCB013739 — INCB013739 50 mg QD tablet
  Arms: Treatment C - INCB013739 & Metformin
Drug: INCB013739 — INCB013739 100 mg QD tablet
  Arms: Treatment D - INCB013739 & Metformin
Drug: INCB013739 — INCB013739 200 mg QD
  Arms: Treatment E - INCB013739 & Metformin
Drug: Placebo comparator matching INCB013739 — Orally once daily tablet
  Arms: Treatment F - Placebo
Drug: Metformin
  Arms: Treatment A - INCB013739 & Metformin; Treatment B - INCB013739 & Metformin; Treatment C - INCB013739 & Metformin; Treatment D - INCB013739 & Metformin; Treatment E - INCB013739 & Metformin

SUMMARY:
Determine the effect of treatment with INCB013739 administered as an 'add-on' to metformin therapy in type 2 diabetic subjects on safety and tolerability and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Type 2 Diabetes
* Stable dose of metformin for more than 8 weeks

Exclusion Criteria:

* Subjects with Addison's disease or Cushing's Syndrome
* Type 1 diabetes mellitus or secondary forms of diabetes
* Subjects with uncontrolled thyroid disease
* History of renal impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in hemoglobin A1c (HbA1c) | Baseline and Week 12 (or early termination study visit)

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in fasting plasma glucose (FPG). | Baseline and Week 12 (or early termination study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Williams, MD, Study Director — Incyte Corporation
Locations (62):
- United States (57):
  - Birmingham, Alabama
  - Artesia, California
  - Calabasas, California
  - Fresno, California
  - Los Angeles, California
  - Los Gatos, California
  - Santa Ana, California
  - Colorado Springs, Colorado
  - Chiefland, Florida
  - Hollywood, Florida
  - Longwood, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Dunwoody, Georgia
  - Rome, Georgia
  - Belleville, Illinois
  - Shawnee Mission, Kansas
  - Bangor, Maine
  - Columbia, Maryland
  - Sterling Heights, Michigan
  - Florissant, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - New York, New York
  - Springfield Gardens, New York
  - West Seneca, New York
  - Calabash, North Carolina
  - Mooresville, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Norton, Ohio
  - Norman, Oklahoma
  - Altoona, Pennsylvania
  - Harleysville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Sellersville, Pennsylvania
  - Greenville, South Carolina
  - North Myrtle Beach, South Carolina
  - Spartanburg, South Carolina
  - Bristol, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Georgetown, Texas
  - Houston, Texas
  - Midland, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Waco, Texas
  - Burke, Virginia
  - Hampton, Virginia
  - Milwaukee, Wisconsin
- Puerto Rico (5):
  - Carolina
  - Fajardo
  - Ponce
  - Río Grande
  - San Juan

REFERENCES:
- [Derived] Rosenstock J, Banarer S, Fonseca VA, Inzucchi SE, Sun W, Yao W, Hollis G, Flores R, Levy R, Williams WV, Seckl JR, Huber R; INCB13739-202 Principal Investigators. The 11-beta-hydroxysteroid dehydrogenase type 1 inhibitor INCB13739 improves hyperglycemia in patients with type 2 diabetes inadequately controlled by metformin monotherapy. Diabetes Care. 2010 Jul;33(7):1516-22. doi: 10.2337/dc09-2315. Epub 2010 Apr 22. PMID 20413513